CLINICAL TRIAL: NCT05399654
Title: A Phase 1/2, Open Label, Dose Escalation and Expansion Study of TAC-001 in Patients With Select Advanced or Metastatic Solid Tumors
Brief Title: A Dose Escalation and Expansion Study of TAC-001 in Patients With Select Advanced or Metastatic Solid Tumors
Acronym: INCLINE-101
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tallac Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCLINE-101
Record Dates: First submitted 2022-05-19; First posted 2022-06-01 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAC-001 Single-Agent Dose-Escalation Cohorts (Experimental)
  Interventions: Drug: TAC-001

INTERVENTIONS:
Drug: TAC-001 — TAC-001 is a Toll-like Receptor Agonist Antibody Conjugate (TRAAC)

SUMMARY:
INCLINE-101 is an open label, multicenter Phase 1/2 study designed to evaluate safety, pharmacokinetics (PK), and preliminary anti-tumor activity of TAC-001 administered intravenously.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically-documented solid tumors.
2. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
3. Demonstrate adequate organ function.

Exclusion Criteria:

1. Prior history of or active malignant disease other than that being treated in this study.
2. Known brain metastases or cranial epidural disease.
3. A known hypersensitivity to the components of the study therapy or its' analogs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2026-05-19 (Estimated)

PRIMARY OUTCOMES:
Dose-Escalation Stage: RP2D for TAC-001 | 2-years
  To identify the recommended dose phase 2 dose (RP2D) for further evaluation of TAC-001 when administered as monotherapy in subjects with advanced or metastatic solid tumors
Dose Expansion: Characterization of ORR for TAC-001 | 2 years
  To evaluate preliminary efficacy of TAC-001 by estimating the overall response rate (ORR; combined complete response [CR] and partial response [PR]) as assessed by the Investigator per RECIST 1.1 and iRECIST
Dose Expansion: Characterization of duration of response for TAC-001 | 2 years
  To evaluate preliminary efficacy of TAC-001 by estimating the duration of response as assessed by the Investigator per RECIST 1.1 and iRECIST
Dose Expansion: Characterization of clinical benefit rate for TAC-001 | 2 years
  To evaluate preliminary efficacy of TAC-001 by estimating the clinical benefit rate as assessed by the Investigator per RECIST 1.1 and iRECIST

SECONDARY OUTCOMES:
Incidence and Severity of Nonserious Adverse Events (AEs) and Serious Adverse Events (SAEs) | 2 years
  To evaluate the safety of TAC-001 monotherapy through the evaluation of incidence and severity of nonserious AEs and SAEs, including immune-related adverse events (irAEs), as graded by investigators according to CTCAE version 5.0
Maximum Plasma Concentration (Cmax) | 2 years
  To evaluate the Cmax of TAC-001 monotherapy
Maximum Plasma Concentration (Tmax) | 2 years
  To evaluate the Tmax of TAC-001 monotherapy
Area Under the Plasma Concentration-Time Curve (AUC) | 2 years
  To evaluate the AUC of TAC-001 monotherapy
Terminal Half-Life | 2 years
  To evaluate the terminal half-life of TAC-001 monotherapy
Clearance of TAC-001 | 2 years
  To evaluate the drug clearance of TAC-001 monotherapy
Evaluation of immunogenicity of TAC-001 | 2 years
  Incidence of antidrug antibodies (ADA) against TAC-001

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - University of Southern California (USC), Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Sarah Cannon Research Institute (SCRI)- Denver, Denver, Colorado
  - AdventHealth Cancer Institute, Orlando, Florida
  - Sarah Cannon Research Institute (SCRI)- Florida Cancer Specialists and Research Institute, LLC, Orlando, Florida
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Weill Cornell Medicine- NYU Clinical Cancer Center, New York, New York
  - West Cancer Center & Research Institute, Germantown, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, Irving, Texas
  - NEXT Oncology- Virginia, Fairfax, Virginia
- Clinical Site, Nedlands, Western Australia, Australia